CLINICAL TRIAL: NCT01723098
Title: Effect of Supervised Exercise Program on Cardiovascular Function and Structure in Pregnant Women. Randomized Controlled Trial
Brief Title: Effect of Regular Exercise on Maternal Cardiovascular System During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD Student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Maternal cardiovascular system
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-03

CONDITIONS: Pregnancy
Keywords: Pregnancy, cardiovascular system, physical exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Sedentary pregnant women
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60 of maximal heart rate. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate.
  Arms: Exercise group

SUMMARY:
The main aim of this study was to analysed the security of a supervised exercise program on maternal cardiovascular system and assess the positive effects of this program on maternal cardiovascular function and structure

DETAILED DESCRIPTION:
During pregnancy, the effectiveness of cardiovascular system is necessary to the growth and development of the baby, however many changes in it occur during this period.

Physical exercise has shown to have a positive effect on cardiovascular structure and function in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Fuenlabrada and Hospital Universitario Severo Ochoa (Madrid).

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from cardiovascular function at the end of pregnancy: Stroke volume | Weeks 20 and 34
  Data were collected in second and third trimester
Change from cardiovascular structure at the end of the pregnancy | Weeks 20 and 34
  Data were collected in second and third trimester

SECONDARY OUTCOMES:
Maternal and fetal pregnancy outcomes | During pregnancy. At the moment of delivery.
  Gestational age, type of delivery, duration of labor, maternal weight gain, birth weight, size and head circumference of new born, pH of umbilical cord, Apgar Score.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Madrid, Spain